CLINICAL TRIAL: NCT05209659
Title: Applying Pain Adaptability to Manual Therapy Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Youngstown State University (Other)
Responsible Party: Principal Investigator, Damian Keter, Principial Investigator, PhD Candidate, Youngstown State University
Other Study IDs: 290
Record Dates: First submitted 2022-01-10; First posted 2022-01-26 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Musculoskeletal Manipulations; Low Back Pain
Keywords: Pan Adaptability
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low Back Pain: Pragmatic Mobilization The pragmatically applied non-thrust manipulation will be based on the original concepts outlined by Maitland and will of consist of passive, low velocity, oscillatory movements within the physiological range of the joint, applied to the comparable spinal level of the patient (defined as the spinal level that reproduced the patient's familiar pain). The techniques will be modified based on clinician assessment and patient feedback and consist of Grade I through Grade IV movements. Since the pragmatic approach is clinician-driven, no time limit will be placed on the application and the number of mobilizations used will depend on the patient feedback (the exact definition of a pragmatic treatment)
  Interventions: Other: Pragmatic Mobilization

INTERVENTIONS:
Other: Pragmatic Mobilization — The techniques will of consist of passive, low velocity, oscillatory movements within the physiological range of the joint, applied to the comparable spinal level of the patient (defined as the spinal level that reproduced the patient's familiar pain). The techniques will be modified based on clinician assessment and patient feedback and consist of Grade I through Grade IV movements. Common techniques used may include unilateral posterior-anterior movements, central posterior-anterior movements, and sidelying rotations (without thrust). Since the pragmatic approach is clinician-driven, no time limit will be placed on the application and the number of mobilizations used will depend on the patient feedback (the exact definition of a pragmatic treatment). Patients will be seen for 4 visits.
  Other Name: Non-thrust manipulation (pragmatically applied)
  Other Names: Mobilization; Mobilisation

SUMMARY:
Mechanism research has identified pain adaptive and non-adaptive phenotypes by documenting the response to an ice immersion bath. Pain adaptive individuals exhibited a rapid response to cold and a rapid resolution of symptoms with continued exposure. Non-pain adaptive individuals had the opposite. Pain-adaptive individuals have the endogenous (internal) capacity to self-modulate pain therefore may pursue active self management techniques, whereas non-pain adaptive phenotypes may be more prone to use of external mechanisms (e.g., analgesic medications) for pain relief. A pain adaptive individual is likely to benefit from all forms of conservative active or passive pain modulatory treatments and is expected to have a favorable prognosis. Although this finding is useful, ice bath immersion is an impractical assessment for clinical practice, leaving clinicians with the inability to identify pain adaptive individuals.

Emerging evidence indicates that an associative clinical response associated with an early within session (during the first visit) and between session (from the first to the second visit) during a posterior to anterior mobilization, identifies individuals who have a favorable prognosis with spinal pain. While neurophysiological basis for the analgesic effect of manual therapy has been proposed to date no one has investigated if the associative clinical response is purely another way of identifying pain adaptive or non-pain adaptive individuals. If a within-session or between-session response is associated with the pain adaptive mechanism found during an ice-bath immersion, clinicians could adopt the clinical evaluation technique and improve their ability to identify proper patients for management. The investigators will evaluate the relationship between the pain adaptive mechanistic response from ice-bath immersion and the associative clinical response that occurs during a PA mobilization of the spine.

DETAILED DESCRIPTION:
This proof-of-concept study uses an observational design to assess correlation between the below stated factors. This study design has been recommended in analgesic management in investigating novel mechanistic relationships. A convenience sample will be recruited from outpatient orthopedic clinics and University sites across a geographically diverse segment of the United States. Individuals will be educated on the purpose and risks of the study via informed consent and will determine if they would like to participate. An a priori power analysis was performed at the .05 significance level with a projected correlation of (.60) and a sample size of 28 participants was recommended to achieve 80 percent power. Given the single session design with virtual/electronic follow up a low dropout rate related to compliance is anticipated. Given the noxious application and the ability to terminate session if requested, along with aforementioned, a total drop-out rate of 10% will be anticipated. A sample size of 32 will be utilized in an attempt to obtain 28 participants.

Data collection will be completed by investigators and/or clinicians whom have been trained directly by investigators on the research protocol or by the research team.

Following consent, the individuals will follow the protocol below:

1. Baseline patient reported measurements will be obtained including McGill Pain Questionnaire, Fear Avoidance Belief Questionnaire, Modified Oswestry Low Back Pain Disability Questionnaire, Expectations of Treatment Scale, Hospital Anxiety and Depression Scale, Fatigue Severity Scale, Numeric Pain Rating Scale (NPRS) (current, best, and worst)
2. Baseline Demographics which have shown prognostic value

   1. Age
   2. Gender
   3. Symptom Duration
   4. Joint(s) involved
   5. Presence of referred leg pain
3. Baseline Objective measures will be obtained including:

   1. Active Range of Motion at lumbar spine and Coxofemoral joint
   2. Neuromuscular Screening (Reflexes, light touch sensation L3-S1, neural testing)
   3. Cardiopulmonary screening (Blood pressure, heart rate, pulse-oximetry, AAA)
   4. Joint mobility at lumbosacral spine via Posterior -> Anterior (PA) mobilizations performed central and unilateral; Assess for comparable sign, If present progress to below
   5. Pain modulation/adaptability assessment - Protocol outlined below:
   6. Application of non-thrust Central or Unilateral PA mobilization application as chosen by the clinician in a pragmatic manner to address patients comparable sign.

      * Technique, grade, time, and location to be recorded
      * Pain (NPRS) to be graded continuously throughout the technique and recorded

   Pain Adaptability/Modulation assessment:

   Throughout the experiment, the participants will sit comfortably in a chair with arms rested on the arm rests and legs testing on the floor. The room temperature will be controlled at 21-23 deg C. Participants will be assured that cold stimulation will not cause any physical damage to their body, and are allowed to withdraw from the experiments at any time.

   Cold pressor pain
   * A bucket of ice and water, a temperature of 1.0C to 4.0C will be maintained by stirring regularly to prevent an increase of water temperature surrounding the hand.
   * Participants will submerge their left hand to 5cm above the wrist with their palm facing down. They will be encouraged to keep their hand in the water for 5 minutes. If they find the pain becoming intolerable, they can withdraw their hand immediately.
   * Pain intensity - During the cold stimulation, participants will be asked to rate the intensity of pain continuously using a 0 to 10 NPRS (0 = no pain at all; 10 = worst pain possible).
   * McGill Pain Questionnaire (MPQ) - will be completed after cold stimulation. The MPQ is designed to provide qualitative and quantitative measures of pain that can be examined statistically. The MPQ consists of 4 major classes of word descriptors (sensory, affective, evaluative, and miscellaneous) for participants to specify subjective pain experience.
   * Pressure pain threshold (PPT) - An electronic pressure algometer (Pain Test FPX 25) with a probe area of 1 cm squared will be used. Participants will indicate when the pressure stimulus becomes just painful. PPT's will be determined by averaging 3 assessments taken at 1-minute intervals. It will take 2 to 3 minutes to complete the PPT tests, which will lead to some participants undertaking a 6-minute cold stimulation test.
   * Sensory assessment - All PPT assessments will be tested at 3 sites: bilateral extensor carpi radialis, at 3 cm distal to the lateral end of the cubic crease on the elbow, and on the right soleus at 8 cm proximal to medial malleolus.
   * All PPT Assessments will be performed before, during (3 minutes after the initiation of cold stimulation), and 20 minutes post termination of Cold Stimulation.
4. 2-week follow up via phone call, text message, email, or virtual meeting to assess NPRS and GROC.

ELIGIBILITY:
Inclusion Criteria:

* History of lumbar spine pain in the past 12 months
* Ability to reproduce low back discomfort with PA mobilization

Exclusion Criteria:

* Demonstration of any signs of upper motor neuron lesion including unexplained loss of function of bowel/bladder, unexplained gait changes, pathologic hyper-reflexia.
* Diagnosis which contradicts the application of prolonged cold including but not limited to severe vascular disease, open wounds/sores on involved extremity.
* Diagnosis which contradicts the application of joint mobilizations including but not limited to instability, inflammatory conditions, severe osteoporosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals whom fit inclusion/exclusion criteria will be recruited from outpatient orthopedic clinics via convenience sample as well as recruited from university and community sites across a geographically diverse segment of the United States.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-12-17 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | collected at baseline and continuously during 5 minute cold pressor test: 2-week follow up via phone call, text message, email, or virtual meeting
  Numeric Pain Rating Scale is a self-reported pain scale which has demonstrated validity and reliability in dealing with multiple pain complaints including chronic spine pain. The scale ranges from 0 to 10 with 0 indicating no perceived pain and 10 indicating maximum perceived pain possible. Aminimally clinically importance difference (MCID) of 1 to 1.7 points or 30% improvement has been suggested.
Global Rating of Change | collected at 2-week follow up via phone call, text message, email, or virtual meeting
  The Global Rating of Change scale is a self-reported scale ranging from -7 (a very great deal worse) to +7 (a very great deal better) with a score of 0 indicating no change from baseline. This scale has demonstrated reliability and validity in assessment of self-reported improvement in the physical therapy profession. Psychometric assessments of this tool have been somewhat limited as it is often utilized as the criterion measure in the assessment of other instruments. A MCID of 2-2.5 points has been suggested.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Learman, PhD, Study Chair — Professor, Department of Graduate Studies in Health and Rehabilitation Sciences, Youngstown State University, Youngstown, Ohio; Severine Van Slambrouck, PhD, Study Director — IRB Director, Youngstown State University, Youngstown, Ohio; Damian L Keter, Principal Investigator — Student, Youngstown State University
Locations (3):
- United States (3):
  - The Therapy Institute, Haslett, Michigan
  - Old Bridge Spine and Wellness, Old Bridge, New Jersey
  - Tri County Physical Therapy Institute, Canfield, Ohio